CLINICAL TRIAL: NCT05649501
Title: Effects of Proprioceptive Neuromuscular Facilitation on Selective Motor Control of Lower Extremity and Balance in Children With Cerebral Palsy
Brief Title: Effect of PNF on Selective Motor Control and Balance in CP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC/22/0725 Misbah Tahir
Record Dates: First submitted 2022-12-06; First posted 2022-12-14 (Actual); Last update posted 2023-04-03 (Actual); Status verified 2023-03

CONDITIONS: CP (Cerebral Palsy)
Keywords: Proprioceptive neuromuscular techniques; Selective voluntary motor control; Balance
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Randomized
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- proprioceptive neuromuscular facilitation techniques (Experimental): Experimental group will receive proprioceptive neuromuscular facilitation stretching which include hold-relax and contract-relax for 6 sec hold, 10 repetitions and 2 min rest in between, for 5 day/week for 4 weeks along with conventional physical therapy.
  Interventions: Other: Proprioceptive neuromuscular facilitation techniques.
- traditional physical therapy (Active Comparator): this group will receive conventional therapy (ROMs, stretching, strengthening).
  Interventions: Other: Proprioceptive neuromuscular facilitation techniques.; Other: Traditional physical therapy

INTERVENTIONS:
Other: Proprioceptive neuromuscular facilitation techniques. — Proprioceptive neuromuscular facilitation stretching which include hold-relax and contract-relax for 6 sec hold, 10 repetitions and 2 min rest in between, for 5 day/week for 4 weeks along with conventional treatment for 40 minutes.
Other: Traditional physical therapy — Conventional therapy (ROMs, stretching, strengthening) of lower limbs for 40 minutes.
  Arms: traditional physical therapy

SUMMARY:
Cerebral palsy is attributed to non-progressive disturbances that occurred in the developing infant brain or fetal characterized by abnormalities of muscle tone, movement and motor skills. PNF technique is thought to have an impact on voluntary motor control and balance through stimulation of proprioceptors, so the aim of this study is to determine the effects of proprioceptive neuromuscular facilitation technique on selective motor control and balance on children with cerebral palsy.

DETAILED DESCRIPTION:
A case study was conducted in 2021 to determine the effects of PNF training for improving lower limb coordination in 7 years old cerebral palsy child. After the intervention, significant improvement is seen in gait parameters, balance, and gross motor functional classification score.

A case report was conducted in 2020, to determine the effectiveness of PNF technique in improving lower extremity function in spastic diplegic cerebral palsied adolescent. Patient was treated with tone inhibitory and movement facilitatory techniques. There was significant change in balance and lower extremity function before and after the treatment.

There are multiple impairments in spastic cerebral palsy children; the inability to perform purposeful voluntary movements is a critical factor in determining functional ability of children. Since selective voluntary motor control is an important factor that must be achieved in cerebral palsy children, PNF may be considered as a technique to gain selective voluntary control and balance proving an important intervention for cerebral palsy children.

ELIGIBILITY:
Inclusion Criteria:

* Children diagnosed as spastic diplegic cerebral palsy
* Age between 5-12 years and both genders.
* Gross motor function level II and III according to gross motor functional classification scale (GMFCS).
* Spasticity range between 1 and 1+ grade according to modified ashworth scale
* Children who are able to follow simple verbal instructions

Exclusion Criteria:

* Children with uncontrolled epilepsy
* Children who show no cooperation
* Children receiving botulinum toxin injections or surgery no earlier than 6 months before project starts.
* Subjects with presence of shortening or deformities of lower limb

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 26 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2023-01-15 (Actual); Study Completion 2023-01-15 (Actual)

PRIMARY OUTCOMES:
Pediatric Berg Balance Scale | last one week
  The Pediatric Balance Scale (PBS), a modification of Berg's Balance Scale, was developed as a balance measure for school-age children with mild to moderate motor impairments. It has 14 items with score 0-4. The intra-class correlation coefficient (ICC) is 0.998 (18).

SECONDARY OUTCOMES:
Selective control assessment of lower extremity (SCALE) | last one week
  The SCALE tool was designed for clinical administration and scoring by healthcare professionals, to be used in less than 15 minutes without specialized equipment. Hip, knee, ankle, subtalar, and toe joints are assessed bilaterally. One representative reciprocal movement that varies from the mass flexor/extensor patterns is chosen to assess SVMC for each joint. Total score is 10 for each limb. Intra-class correlation coefficient ranges from 0.88 to 0.91 (19).

CONTACTS AND LOCATIONS:
Overall Officials: Shabana Ashraf, Masters, Principal Investigator — Riphah International University
Locations (1):
- Pakistan Society for Rehabilitation of the Disabled (PSRD), Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mutch L, Alberman E, Hagberg B, Kodama K, Perat MV. Cerebral palsy epidemiology: where are we now and where are we going? Dev Med Child Neurol. 1992 Jun;34(6):547-51. doi: 10.1111/j.1469-8749.1992.tb11479.x. No abstract available. PMID 1612216
- [Background] Bax M, Goldstein M, Rosenbaum P, Leviton A, Paneth N, Dan B, Jacobsson B, Damiano D; Executive Committee for the Definition of Cerebral Palsy. Proposed definition and classification of cerebral palsy, April 2005. Dev Med Child Neurol. 2005 Aug;47(8):571-6. doi: 10.1017/s001216220500112x. PMID 16108461
- [Background] Rosenbaum P, Paneth N, Leviton A, Goldstein M, Bax M, Damiano D, Dan B, Jacobsson B. A report: the definition and classification of cerebral palsy April 2006. Dev Med Child Neurol Suppl. 2007 Feb;109:8-14. PMID 17370477
- [Background] Tang-Wai R, Webster RI, Shevell MI. A clinical and etiologic profile of spastic diplegia. Pediatr Neurol. 2006 Mar;34(3):212-8. doi: 10.1016/j.pediatrneurol.2005.08.027. PMID 16504791
- [Background] 15. Akalan E, Ertürk G, Önerge K, Evrendirek H, Karaca G. Investigation of the Relationship Between Selective Voluntary Motor Control and Static Balance in Cerebral Palsy. 2019.
- [Background] Franjoine MR, Darr N, Held SL, Kott K, Young BL. The performance of children developing typically on the pediatric balance scale. Pediatr Phys Ther. 2010 Winter;22(4):350-9. doi: 10.1097/PEP.0b013e3181f9d5eb. PMID 21068635
- [Background] Balzer J, Marsico P, Mitteregger E, van der Linden ML, Mercer TH, van Hedel HJ. Construct validity and reliability of the Selective Control Assessment of the Lower Extremity in children with cerebral palsy. Dev Med Child Neurol. 2016 Feb;58(2):167-72. doi: 10.1111/dmcn.12805. Epub 2015 May 20. PMID 25991061